CLINICAL TRIAL: NCT00866203
Title: A Prospective, Randomized, Multicenter Trial Comparing a Modified HDS Therapy Supported by PBPC Transplant With Additional 4 Courses of Front-Line Therapy in Adult Aggressive NHL With PR After Short Course of Up-Front Chemotherapy
Brief Title: HDS Plus PBPC Transplant Vs 4 More Courses of FrontLine Therapy in Pts With Aggressive NHL in PR After Induction Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: sponsor, Gruppo Italiano Studio Linfomi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LA05
Record Dates: First submitted 2007-03-13; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: High-Grade Lymphomas
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HDS (Experimental): modified high dose sequential therapy
  Interventions: Drug: HDS vs ProMECE/CytaBOM
- ProMECE/CytaBOM (Active Comparator): four additional courses of standard ProMECE/CytaBOM
  Interventions: Drug: HDS vs ProMECE/CytaBOM

INTERVENTIONS:
Drug: HDS vs ProMECE/CytaBOM

SUMMARY:
The study is planned to compare the outcome of aggressive NHL patients in partial remission after four courses of front-line therapy, randomly assigned to receive either additional four courses of the same regimen or a modified HDS program.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, untreated patients with histologically documented aggressive lymphoma;
* Age between 18 and 65 years;
* Clinical stage at diagnosis: I A bulky - IV B;
* Reduction of tumoral masses, after four courses of induction therapy, between 50 and 75%;
* Serum negativity for HIV, HbsAg and HCV;
* ECOG performance status 0 through 4;
* Adequate bone marrow function;
* Adequate renal and hepatic functions;
* Left ventricular ejection fraction (LVEF) > 50%;
* No previous malignant disease;
* No previous chemo-radiotherapy;
* No cerebral or CNS involvement, assessed by clinical history, physical examination and CSF examination through lumbar puncture;
* Written informed consent given at time of randomization.

Exclusion Criteria:

* Clinical stage I no bulky, or CS IIA-B with less than three sites of disease involved;
* Patients with CR, unconfirmed complete remission (uCR), very good PR (>75%) and clinical response less than 50%, as defined by Cheson et al., following four courses of induction therapy;
* Tumor involvement of CNS (except patients with peridural masses without liquor involvement , who can be enrolled in this study);
* Indolent lymphoma transformed in more aggressive histologic type, even if never previously treated;
* Aggressive non-Hodgkin's lymphoma in pre-transplanted patient;
* Clinically significant secondary cardiovascular disease e.g. uncontrolled hypertension, (resting diastolic blood pressure > 115 mmHg), uncontrolled multifocal cardiac arrhythmias, symptomatic angina pectoris or congestive cardiac failure NYHA class III-IV;
* Left ventricular ejection fraction (LVEF) < 50%;
* Evidence of any severe active acute or chronic infection;
* Concurrent malignancy of history of other malignancy, except basal cell carcinoma of the skin (BCC) and in situ cervical carcinoma (CIN);
* myelodisplastic syndrome;
* HbsAg, HIV-positive, or HCV-RNA-positive patients;
* Patient with psychiatric, or any disorder that compromises ability to give truly informed consent for participation in this study;
* Pregnant woman; potential child-bearing women can be enrolled if adequate contraceptive precautions are used before entering this trial and for the duration of the trial;
* Concerns for patient's compliance with the protocol procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2000-10; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
remission duration | end of treatment
overall survival | study end
event-free survival | study end
freedom-from progression | study end

SECONDARY OUTCOMES:
feasibility and toxicity | end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Di Renzo, MD, Principal Investigator — GISL; Massimo Federico, MD, Study Chair — GISL; Maura Brugiatelli, MD, Study Chair — GISL; Mario Petrini, MD, Study Chair — GISL; Paolo G Gobbi, MD, Study Chair — GISL
Locations (1):
- GISL Trial Office, Modena, Italy